CLINICAL TRIAL: NCT00702533
Title: A New Method for Determining Gastric Acid Output Using a Wireless Capsule
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080138; 08-DK-0138
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-06

CONDITIONS: Gastric Acid Secretory Disorders
Keywords: Gastric Acid Output; Hyper/Hyposecretion; Gastric Analysis; Gastric pH; SmartPill; Natural History; Gastric Secretion; Healthy Volunteer; HV
MeSH Terms: interventions — Pentagastrin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy volunteers between 18 and 60 years of age
  Interventions: Device: Pentagastrin Injection BP
- patients with gastric acid secretory disorders: 18 years of age who have been diagnosed with Zollinger-Ellison Syndrome or acid hypersecretion.
  Interventions: Device: Pentagastrin Injection BP; Drug: Pentagastrin

INTERVENTIONS:
Device: Pentagastrin Injection BP
Drug: Pentagastrin
  Groups: patients with gastric acid secretory disorders

SUMMARY:
Background:

- Acid-related gastrointestinal disorders are numerous and may require chronic treatment and maintenance, but they are often difficult to diagnose and treat. Gastric analysis is a critical tool for diagnosing and treating acid-related disorders; however, at present it requires a technically difficult procedure, using a nasogastric tube, that is costly, invasive, and uncomfortable. Recently a new tool, the SmartPill, has been developed that can measure acid levels, temperature, and pressure throughout the stomach, small intestine, and colon by swallowing a small capsule. Researchers are interested in comparing current methods of measuring stomach acid with the SmartPill by studying both healthy volunteers and individuals with acid-related gastrointestinal disorders.

Objectives:

- To evaluate the usefulness and accuracy of the SmartPill for gastric analysis, compared with current procedures.

Eligibility:

* Phase 1A/1B: Healthy volunteers between 18 and 60 years of age.
* Phase 2: Individuals at least 18 years of age who have been diagnosed with Zollinger-Ellison Syndrome or acid hypersecretion.
* Phase 3: Individuals at least 18 years of age who have been diagnosed with refractory gastroesophageal reflux disease, peptic ulcer disease, or idiopathic gastric hypersecretion.

Design:

* This study involves a screening visit, a 3-day inpatient study visit, and possible additional outpatient visits.
* Participants will be screened with a medical history and physical examination, as well as blood and urine samples.
* Phase 1A/1B: Participants will have a 3-day inpatient study visit with the following procedures:
* Imaging study of the stomach (simultaneous gastric emptying scintigraphy), followed by a special diet for the next day s test.
* Gastric analysis using a nasogastric tube to collect stomach acid secretions.
* SmartPill study, in which participants will ingest a SmartPill and wear a monitor for 24 to 48 hours to collect readings.
* Participants in Phase 1A will have a second outpatient SmartPill study 7 days after the first SmartPill study. Participants in Phase 1B will not have the second SmartPill study.
* Phase 2 and Phase 3: Participants will have a 3-day inpatient study visit with the following procedures:
* Imaging study of the stomach (simultaneous gastric emptying scintigraphy), followed by a special diet for the next day s test.
* Gastric analysis using a nasogastric tube to collect stomach acid secretions.
* SmartPill study, in which participants will ingest a SmartPill and wear a monitor for 24 to 48 hours to collect readings.
* Phase 2 and 3 participants will have outpatient study visits only if directed by the study researchers....

DETAILED DESCRIPTION:
Acid related disorders are numerous and often require chronic treatment and maintenance. Many of these diseases are without symptoms and therefore difficult to diagnose and treat. Gastric analysis is the quantitative measurement of gastric acid output and is a critical tool for the diagnosis of acid related disorders and the ongoing assessment of therapy response. At present gastric analysis requires a technically difficult procedure, using gastric aspiration through a nasogastric tube, that is costly, invasive, and uncomfortable for patients. Recently there is introduction of the SmartPill, which is a disposable pill that measures pH, temperature, and pressure throughout the GI tract. We propose a pilot study to validate a new method of gastric analysis with the ingestion of the SmartPill with a meal of a known buffering capacity to measure both the acidity and quantity of acid output in the stomach. We will validate this method by comparing it to the accepted gastric aspiration method under maximally stimulated conditions. We will study healthy volunteers for the validation phase and then study patients with known acid related disorders to assess its usefulness in patients. Interested subjects will report to the NIH outpatient gastrointestinal clinic for evaluation to be followed by a 3 day in-patient admission and 2 subsequent clinic visits. Subjects will have gastric analysis of basal, meal stimulated, and pharmacologically stimulated rates with both the conventional and study methods. Outcomes will include a quantitative measurement of gastric acid output in unit time, normal meal stimulated acid output values in healthy volunteers and patients with acid related disorders, and the assessment of acid suppression in patients treated with a variety of anti-secretory medications.

ELIGIBILITY:
* CURRENTLY ONLY RECRUITING Patients with Zollinger Ellison Syndrome and Hypersecretion AND Patients with Refractory GERD, Peptic ulcer disease, Idiopathic Gastric Hypersecretion

Phase II, Use in Patients with Zollinger Ellison Syndrome and Hypersecretion

INCLUSION:

* Zollinger-Ellison syndrome (ZES) as diagnosed by one of the following criteria: histologic confirmation of gastrinoma, positive provocative testing with secretin (an increase of >200 pg/mL postinjection), gastric acid hypersecretion (BAO > 15) in the presence of hypergastrinemia (fasting serum gastrin > 99)
* Multiple endocrine neoplasia type-I (MEN1) with suspicion of ZES (hypergastrinemia) undergoing evaluation. MEN-I with ZES
* Hypergastrinemia (serum gastrin > 99)

Patients must meet at least 1 of the above inclusion criteria and the following:

* Ages equal to or greater than 18 years
* Male, females, all ethnicities

EXCLUSION:

* History of gastric surgery (gastrectomy, pyloroplasty)
* Use of bowel motility medications such as, but not limited to, Reglan, Immodium, and Lomotil
* Contraindication to SmartPill: history of gastric bezoar, disorders of swallowing, suspected strictures, fistulas, or physiological GI obstruction, GI surgery within the past three months, severe dysphagia to food or pills, Crohn s Disease or diverticulitis, a subject who uses an implanted or portable electro-mechanical medical device such as a cardiac pacemaker or infusion pump
* Pregnancy and breastfeeding. Females of childbearing potential must be on an acceptable means of birth control and no intercourse in 2 weeks prior to study enrollment.
* Lactose intolerance or inability to drink standard meal of Ensure Plus
* Estabished diagnosis of gastroparesis
* Significant systemic or major illnesses including, but not limited to, stroke, congestive heart failure, renal failure (creatinine clearance < 50 ml/min), organ transplantation, angina pectoris, active malignancy, and autonomic neuropathy
* Unstable psychiatric conditions, untreated or uncontrolled depression or generalized anxiety disorder, substance abuse within the past year, in order to prevent feeling of being uncomfortable or to prevent lack of follow-up
* Use of not-steroidal anti-inflammatory drugs for 2 weeks prior to study enrollment

Phase IIIA, Use in Patients with Refractory GERD, Peptic ulcer disease, Idiopathic Gastric Hypersecretion

INCLUSION:

* Gastric acid hypersecretion (BAO>15 mEq/hr)
* Conditions with gastric acid hypersecretion including, but not limited to, patients with systemic mastocytosis (SM)
* Refractory GERD (patients with persistant symptoms despite being on standard medical therapy), PUD, and suspected idiopathic gastric hypersecretion

Patients must meet at least 1 of the above inclusion criteria and the following:

* Ages equal to or greater than 18 years
* Male, females, all ethnicities

EXCLUSION:

* History of gastric surgery (gastrectomy, pyloroplasty).
* Use of bowel motility medications such as, but not limited to, Reglan, Immodium, and Lomotil
* Contraindication to SmartPill: history of gastric bezoar, disorders of swallowing, suspected strictures, fistulas, or physiological GI obstruction, GI surgery within the past three months, severe dysphagia to food or pills, Crohn s Disease or diverticulitis, a subject who uses an implanted or portable electro-mechanical medical device such as a cardiac pacemaker or infusion pump
* Pregnancy and breastfeeding. Females of childbearing potential must be on an acceptable means of birth control and no intercourse in 2 weeks prior to study enrollment.
* Lactose intolerance or inability to drink standard meal of Ensure Plus
* Established diagnosis of gastroparesis
* Significant systemic or major illnesses including, but not limited to, stroke, congestive heart failure, renal failure (creatinine clearance < 50 ml/min), organ transplantation, angina pectoris, active malignancy, and autonomic neuropathy
* Unstable psychiatric conditions, untreated or uncontrolled depression or generalized anxiety disorders, substance abuse within the past year, in order to prevent feeling of being uncomfortable or to prevent lack of follow-up. Use of non-steroidal anti-inflammatory drugs for 2 weeks prior to study enrollment.

Phase IIIB, Use in Patients with Medication-Controlled: GERD, Peptic ulcer disease, Idiopathic Gastric Hypersecretion

INCLUSION:

-Medication-controlled (patients whose symptoms resolve with medication):GERD, PUD, and suspected idiopathic gastric hypersecretion

Patients must meet the above inclusion criteria and the following

* Ages equal to or greater than 18 years
* Male, females, all ethnicities

EXCLUSION:

* Refractory to medication: GERD (patients with persistant symptoms despite being on standard medical therapy), PUD, and suspected idiopathic gastric hypersecretion
* History of gastric surgery (gastrectomy, pyloroplasty).
* Use of bowel motility medications such as, but not limited to, Reglan, Immodium, and Lomotil
* Contraindication to SmartPill: history of gastric bezoar, disorders of swallowing, suspected strictures, fistulas, or physiological GI obstruction, GI surgery within the past three months, severe dysphagia to food or pills, Crohn s Disease or diverticulitis, a subject who uses an implanted or portable electro-mechanical medical device such as a cardiac pacemaker or infusion pump
* Pregnancy and breastfeeding. Females of childbearing potential must be on an acceptable means of birth control and no intercourse in 2 weeks prior to study enrollment.
* Lactose intolerance or inability to drink standard meal of Ensure Plus
* Established diagnosis of gastroparesis
* Significant systemic or major illnesses including, but not limited to, stroke, congestive heart failure, renal failure (creatinine clearance < 50 ml/min), organ transplantation, angina pectoris, active malignancy, and autonomic neuropathy
* Unstable psychiatric conditions, untreated or uncontrolled depression or genralized anxiety disorders, substance abuse within the past year, in order to prevent feeling of being uncomfortable or to prevent lack of follow-up
* Use of non-steroidal anti-inflammatory drugs for 2 weeks prior to study enrollment

RECRUITMENT IS CLOSED FOR Phase IA/IB, Validation and Establishment of Nomogram in Healthy Volunteers

PHASE IA/IB INCLUSION:

* Healthy volunteers
* Ages 18-60
* Males, females, all ethnicities

PHASE IA/IB EXCLUSION:

* History of gastric or bowel surgery
* Use of bowel motility medications such as, but not limited to, Reglan, Immodium, and Lomotil
* Use of antacid, antisecretory, and anticholinergic medications such as, but not limited to, proton pump inhibitors and histamine 2 receptor antagonists
* Use of non-steroidal anti-inflammatory drugs for 2 weeks prior to study enrollment
* Hypersecretory and hyposecretory related conditions including, but not limited to, pernicious anemia, atrophic gastritis, and Zollinger-Ellison syndrome
* Contraindication to NGT: deviated septum, history of transphenoidal surgery, chronic sinusitis, severe facial trauma (cribriform plate disruption, sustained head trauma, maxillofacial injury, or anterior fossa skull fracture), esophageal stricture, esophageal varices, altered mental status, and impaired airway
* Contraindication to scintigraphy: allergy to sulfa-colloid
* Contraindication to pentagastrin: allergy to pentagastrin, active gastrointestinal bleeding, active peptic ulcer disease, active gallbladder and liver disease, pancreatitis, and bowel obstruction
* Contraindication to SmartPill: history of gastric bezoar, disorders of swallowing, suspected strictures, fistulas, or physiological GI obstruction, GI surgery within the past three months, severe dysphagia to food or pills, Crohns disease or diverticulosis, and implanted or portable electro-mechanical medical device such as a cardiac pacemaker or infusion pump
* Pregnancy and breastfeeding. Females of childbearing potential must be on an acceptable means of birth control and no intercourse in 2 weeks prior to study enrollment.
* Lactose intolerance or inability to drink standard meal of Ensure Plus
* Helicobacter pylori infection
* Gastroparesis
* History of gastroesophageal reflux disease, peptic ulcer disease, irritable bowel syndrome, or inflammatory bowel disease
* Significant systemic or major illnesses including, but not limited to, stroke, cardiovascular disease, hypertension, congestive heart failure, renal failure (creatinine clearance < 50 ml/min), organ transplantation, angina pectoris, active malignancy, diabetes, or autonomic neuropathy
* Unstable psychiatric conditions, depression, generalized anxiety disorder, or substance abuse within the past year, in order to prevent feeling of being uncomfortable or to prevent lack of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with gastric acid secretory disorders
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-06-18

PRIMARY OUTCOMES:
examines the safety and efficacy of disposable, wireless capsule (SmartPill) | until protocol closes
  This study examines the safety and efficacy of disposable, wireless capsule (SmartPill) devices in determining gastric acid output in comparison to current standard gastric aspiration procedures, which are more invasive and inconvenient.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Wank, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shaheen NJ, Hansen RA, Morgan DR, Gangarosa LM, Ringel Y, Thiny MT, Russo MW, Sandler RS. The burden of gastrointestinal and liver diseases, 2006. Am J Gastroenterol. 2006 Sep;101(9):2128-38. doi: 10.1111/j.1572-0241.2006.00723.x. Epub 2006 Jul 18. PMID 16848807
- [Background] Bruley Des Varannes S, Marek L, Humeau B, Lecasble M, Colin R. Gastroesophageal reflux disease in primary care. Prevalence, epidemiology and Quality of Life of patients. Gastroenterol Clin Biol. 2006 Mar;30(3):364-70. doi: 10.1016/s0399-8320(06)73189-x. PMID 16633300
- [Background] El-Serag HB, Aguirre T, Kuebeler M, Sampliner RE. The length of newly diagnosed Barrett's oesophagus and prior use of acid suppressive therapy. Aliment Pharmacol Ther. 2004 Jun 15;19(12):1255-60. doi: 10.1111/j.1365-2036.2004.02006.x. PMID 15191506
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-DK-0138.html